CLINICAL TRIAL: NCT06323642
Title: Role of Probiotics as Adjunct Therapy Along With Standard Care in Decreasing Hospital Stay and Improving Symptoms in Pediatric Patients Admitted With Severe Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Nighat Haider, assisstant professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F.1-1/20ERB/SZABMU/941
Record Dates: First submitted 2024-03-04; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pneumonia; Probiotics
Keywords: pneumonia treatment; probiotics
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Participant
Masking Description: The patients and their parents/attendants will be kept blind to the fact that they are receiving either probiotic or placebo
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): probiotic mixture will be given daily to patients probiotic mixture containing: Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: probiotic containing Lactobacillus rhamnosus GG.
- B (Placebo Comparator): placebo mixture will be given to patients with pneumonia
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: probiotic containing Lactobacillus rhamnosus GG. — probiotic containing Lactobacillus rhamnosus GG will be given daily for 3 days
  Arms: A
Other: placebo — milk as placebo
  Arms: B

SUMMARY:
Probiotics as adjuvant therapy along with standard care can decrease hospital stay and improve symptoms (fever, tachypnea,cough) in pediatric patients admitted with severe pneumonia.

DETAILED DESCRIPTION:
After getting written informed consent from parents/attendants, all patients aged 6 month-2yrs admitted with severe pneumonia in pediatric wards of children hospital, during the study time of 6 month will be recruited.After applying exclusion criteria remaining participants will be included in the study. The study population will be randomized in to two groups, Group A will be given probiotic sachet and group B will be given simple milk as placebo.The patients and their parents/attendants will be kept blind to the fact that they are receiving either probiotic or placebo The probiotic and placebo mixture will be given daily for three days.The patients in both the groups will be followed for the duration of illness until they are either discharged or show any adverse outcomes of pneumonia.Total days of admission will be recoded for patients discharged from hospital.Parents will be asked questions regarding improvement in symptoms like fever on discharge. Duration for Improvement in tachypnea andcough will be noted for all patients. Outcomes will be duration of hospital admission, improvement in fever, tachypnea and cough.All the data collected will be entered and analyzed using SPSS latest version and analysed.

ELIGIBILITY:
Inclusion criteria Patient aged 2month-24months. Both male and female children

Exclusion Criteria:

Patients with severe acute malnutrition Patients with very severe pneumonia Patients with Other concurrent infections Patients having any chronic debilitating condition Children who took probiotics in past 6 months Patient requiring mechanical ventilation

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of days in hospital | 6 month
  hospital stay in patients admitted with severe pneumonia.

SECONDARY OUTCOMES:
Number of days with cough, fever | 6 month
  Improving symptoms in patients admitted with severe pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Nighat Haider, Study Chair — SZABMU
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No